CLINICAL TRIAL: NCT01363128
Title: Phase II Study of the Hyper - CVAD Regimen in Combination With Ofatumumab as Frontline Therapy for Patients With CD-20 Positive Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy and Ofatumumab in Treating Patients With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0708; NCI-2011-01061 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0708 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia; Adult Acute Lymphoblastic Leukemia in Complete Remission; Burkitt Leukemia; Burkitt Lymphoma; CD20 Positive; Childhood Acute Lymphoblastic Leukemia in Complete Remission; Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Methotrexate; merphos; ofatumumab; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (hyper-CVAD, ofatumumab) (Experimental): COURSES 1, 3, 5, 7: Patients receive hyper-CVAD comprising cyclophosphamide IV over 3 hours every 12 hours on days 1-3; doxorubicin hydrochloride IV over 24 hours on day 4; vincristine sulfate IV over 15 minutes on days 4 and 11; and dexamethasone IV over 30 minutes or PO QD on days 1-4 and 11-14. Patients also receive ofatumumab IV over 4-6 hours on days 1 and 11 of courses 1 and 3.
  COURSES 2, 4, 6, 8: Patients receive high-dose methotrexate IV over 2 hours and then over 22 hours on day 1 and cytarabine IV over 2 hours every 12 hours on days 2-3. Patients also receive ofatumumab IV over 4-6 hours on days 1 and 8 of courses 2 and 4.
  Treatment repeats every 21-28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients may receive maintenance therapy for an additional 30 months.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Biological: Ofatumumab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well combination chemotherapy and ofatumumab work in treating patients with acute lymphoblastic leukemia or lymphoblastic lymphoma. Drugs used in chemotherapy, such as cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with ofatumumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving combination chemotherapy together with ofatumumab may be an effective treatment for acute lymphoblastic leukemia or lymphoblastic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical efficacy of the combination of hyper-CVAD (cyclophosphamide, vincristine sulfate, doxorubicin hydrochloride, and dexamethasone) + ofatumumab in patients with newly diagnosed acute lymphoblastic leukemia with any level of CD20 expression: event-free survival; overall response rate; overall survival.

SECONDARY OBJECTIVES:

I. To evaluate the safety of this combination.

OUTLINE:

COURSES 1, 3, 5, 7: Patients receive hyper-CVAD comprising cyclophosphamide intravenously (IV) over 3 hours every 12 hours on days 1-3; doxorubicin hydrochloride IV over 24 hours on day 4; vincristine sulfate IV over 15 minutes on days 4 and 11; and dexamethasone IV over 30 minutes or orally (PO) once daily (QD) on days 1-4 and 11-14. Patients also receive ofatumumab IV over 4-6 hours on days 1 and 11 of courses 1 and 3.

COURSES 2, 4, 6, 8: Patients receive high-dose methotrexate IV over 2 hours and then over 22 hours on day 1 and cytarabine IV over 2 hours every 12 hours on days 2-3. Patients also receive ofatumumab IV over 4-6 hours on days 1 and 8 of courses 2 and 4.

Treatment repeats every 21-28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients may receive maintenance therapy for an additional 30 months.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with newly diagnosed, previously untreated CD-20+ acute lymphoblastic leukemia (ALL), or lymphoblastic lymphoma, Burkitt leukemia/lymphoma or having achieved complete remission (CR) with one course of induction chemotherapy
* Failure to one induction course of chemotherapy (these patients will be analyzed separately)
* Performance status of 0, 1, or 2
* Creatinine less than or equal to 3.0 mg/dL (unless considered tumor related)
* Bilirubin less than or equal to 3.0 mg/dL (unless considered tumor related)
* Adequate cardiac function defined as no clinically significant history of arrhythmia as determined by the principal investigator (PI) and/or the treating physician, history of myocardial infarction (MI) or clinically significant abnormal electrocardiogram (EKG), as determined by the PI and/or the treating physician, within 3 months prior to study enrollment; cardiac function will be assessed by history and physical examination
* No active or co-existing malignancy (other than ALL or lymphoblastic lymphoma) with life expectancy less than 12 months due to that malignancy

Exclusion Criteria:

* Pregnant or nursing women
* Known to be human immunodeficiency virus positive (HIV+)
* Philadelphia chromosome (Ph)+ ALL
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half-lives (calculated by multiplying the reported terminal half-life by 5) or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Positive serology for hepatitis B (HB) defined as a positive test for hepatitis B surface antigen (HBsAg); in addition, if negative for HBsAg but hepatitis B core antibody (HBcAb) positive (regardless of HBsAb status), a HB deoxyribonucleic acid (DNA) test will be performed and if positive the subject will be excluded; consult with a physician experienced in care & management of subjects with hepatitis B to manage/treat subjects who are anti-HBc positive
* Positive serology for hepatitis C (HC) defined as a positive test for hepatitis C antibody (HCAb), in which case reflexively perform a HC radioimmunoblotting assay (RIBA) immunoblot assay on the same sample to confirm the result

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-07-12 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Sasaki K, Kantarjian HM, Morita K, Short NJ, Konopleva M, Jain N, Ravandi F, Garcia-Manero G, Wang S, Khoury JD, Jorgensen JL, Champlin RE, Khouri IF, Kebriaei P, Schroeder HM, Khouri M, Garris R, Takahashi K, O'Brien SM, Jabbour EJ. Hyper-CVAD plus ofatumumab versus hyper-CVAD plus rituximab as frontline therapy in adults with Philadelphia chromosome-negative acute lymphoblastic leukemia: A propensity score analysis. Cancer. 2021 Sep 15;127(18):3381-3389. doi: 10.1002/cncr.33655. Epub 2021 Jun 17. PMID 34138471
- [Derived] Jabbour E, Richard-Carpentier G, Sasaki Y, Konopleva M, Patel K, Roberts K, Gu Z, Wang F, Huang X, Sasaki K, Short NJ, Jain N, Ravandi F, Daver NG, Kadia TM, Alvarado Y, DiNardo CD, Issa GC, Pemmaraju N, Garcia-Manero G, Verstovsek S, Wang S, Khoury JD, Jorgensen J, Champlin R, Khouri I, Kebriaei P, Schroeder H, Khouri M, Mullighan CG, Takahashi K, O'Brien SM, Kantarjian H. Hyper-CVAD regimen in combination with ofatumumab as frontline therapy for adults with Philadelphia chromosome-negative B-cell acute lymphoblastic leukaemia: a single-arm, phase 2 trial. Lancet Haematol. 2020 Jul;7(7):e523-e533. doi: 10.1016/S2352-3026(20)30144-7. PMID 32589978
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2011 to May 2017
Groups:
- Treatment (Hyper-CVAD, Ofatumumab): COURSES 1, 3, 5, 7: Patients receive hyper-CVAD comprising cyclophosphamide IV over 3 hours every 12 hours on days 1-3; doxorubicin hydrochloride IV over 24 hours on day 4; vincristine sulfate IV over 15 minutes on days 4 and 11; and dexamethasone IV over 30 minutes or PO QD on days 1-4 and 11-14. Patients also receive ofatumumab IV over 4-6 hours on days 1 and 11 of courses 1 and 3.
  COURSES 2, 4, 6, 8: Patients receive high-dose methotrexate IV over 2 hours and then over 22 hours on day 1 and cytarabine IV over 2 hours every 12 hours on days 2-3. Patients also receive ofatumumab IV over 4-6 hours on days 1 and 8 of courses 2 and 4.
  Treatment repeats every 21-28 days for 8 courses in the absence of disease progression or unacceptable toxicity. Patients may receive maintenance therapy for an additional 30 months.
  Cyclophosphamide: Given IV
  Cytarabine: Given IV
  Dexamethasone: Given IV or PO
  Doxorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IV
  Ofatumumab: Given IV
  Vincristine Sulfate: Given IV
Period: Overall Study
Arm/Group | Treatment (Hyper-CVAD, Ofatumumab)
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Hyper-CVAD, Ofatumumab)
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 41 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 53
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission (CR)
Description: Complete Remission is Normalization of the peripheral blood and bone marrow with 5% or less blasts in marrow with a granulocyte count of 1 x 109/L or above and a platelet count of 100x 109/L or above. Complete resolution of all sites of extramedullary disease is required for CR.
Time Frame: Up to 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hyper-CVAD, Ofatumumab)
Number analyzed (Participants) | 69
Participants | 68

2. Primary Outcome: 4-Year Overall Survival
Description: Overall Survival is defined as time from date of treatment start until date of death due to any cause or last Follow-up. For continuous data, summary statistics including n, mean, standard deviation, median, minimum and maximum will be computed. The posterior median time to event and it 95% credible interval will be estimated. Kaplan-Meier method, Log rank test and Cox proportional hazards regression modeling will be utilized to analyze survival at 4 years.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hyper-CVAD, Ofatumumab)
Number analyzed (Participants) | 69
Participants | 47

3. Primary Outcome: 4-year Event Free Survival
Description: Event Free Survival defined as the time from the start of therapy to time of primary refractory disease, relapse from CR, death from any cause or last follow-up. Kaplan-Meier method will be utilized to analyze event free survival for the 4 year percent alive and in CR.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Hyper-CVAD, Ofatumumab)
Number analyzed (Participants) | 69
Participants | 41

ADVERSE EVENTS:
Time Frame: Up to 8 years 9 months
Arm/Group | Treatment (Hyper-CVAD, Ofatumumab)
All-Cause Mortality (participants affected / at risk) | 1/69
Serious Adverse Events (participants affected / at risk) | 46/69
Other Adverse Events (participants affected / at risk) | 48/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hyper-CVAD, Ofatumumab) (N=69)
Alanine Aminotransferase Increased (Investigations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cholecyisitis (Hepatobiliary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear Other (Ear and labyrinth disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye Disorders (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 10 (13)
Fever (General disorders) | 7 (8)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 3 (4)
Headache (General disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 30 (59)
Infusion Related Reaction (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 15 (26)
Meningitis (Infections and infestations) | 1 (1)
Muscle Weakness (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasm benign, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous System Disorder (Nervous system disorders) | 1 (2)
Oral Hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 5 (5)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Peripheral Ischemia (Vascular disorders) | 1 (1)
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1)
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 1 (1)
Sepsis (Infections and infestations) | 9 (11)
Sinus Tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 3 (4)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Hyper-CVAD, Ofatumumab) (N=69)
Alanine Aminotransferase Increased (Investigations) | 14 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 11 (21)
Aspartate Aminotransferase Increased (Investigations) | 5 (5)
Blood Bilirubin Increased (Investigations) | 4 (4)
Catheter Related Infection (Infections and infestations) | 4 (5)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Neutropenic Fever (Infections and infestations) | 10 (10)
Fever (General disorders) | 7 (7)
Headache (General disorders) | 7 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (21)
Infection (Infections and infestations) | 8 (10)
Infusion Related Reaction (Investigations) | 12 (13)
Insomnia (Nervous system disorders) | 4 (4)
Oral Mucositis (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 13 (17)
Neutropenia (Investigations) | 19 (57)
Pain in Extremity (General disorders) | 4 (9)
Peripheral Sensory Neuropathy (Nervous system disorders) | 4 (7)
Thrombocytopenia (Investigations) | 17 (45)
Sepsis (Infections and infestations) | 4 (4)
Skin Infection (Infections and infestations) | 4 (4)
Upper Respiratory Infection (Infections and infestations) | 5 (7)
Vomiting (Gastrointestinal disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT01363128/Prot_SAP_000.pdf